CLINICAL TRIAL: NCT05333328
Title: Endocrine Therapies With Ovarian Function Suppression in Premenopausal Node+ Early Breast Cancer With Low Genomic Risk (INTERSTELLAR Trial, KBCSG-25)
Brief Title: OFS in Premenopausal Node+ Breast Cancer With Low Genomic Risk
Acronym: INTERSTELLAR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Collaborators: Seoul National University (Other)
Responsible Party: Principal Investigator, Sung Gwe Ahn, Associated Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1151-002
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Estrogen Receptor Positive Tumor; HER2-negative Breast Cancer; Premenopausal Breast Cancer; Node-positive Breast Cancer
Keywords: Breast Cancer; Estrogen Receptor Positive Tumor; HER2-negative Breast Cancer; Premenopausal Breast Cancer; Node-positive Breast Cancer; Multigene assay; Ovarian-function suppression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: De-escalating treatment as ovarian-function suppression with endocrine treatments alone in ER+HER2- premenopausal women with N1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OFS with endocrine (Experimental): Among ER+HER2- premenopausal patients with N1 who undergoes primary breast surgery, the patients with a genomic low risk using the multigene-assay (OncoFREE®) will be included in this arm.
  Interventions: Drug: Ovarian function suppression with endocrine treatments

INTERVENTIONS:
Drug: Ovarian function suppression with endocrine treatments — * Ovarian function suppression (OFS) with endocrine therapies including either tamoxifen or aromatase-inhibitors will be administered for 5 years.
  * Either goserelin acetate or leuprorelin Acetate is allowed.
  * These patients are able to choose bilateral salpingo-oophorectomy instead of OFS.
  * Chemotherapy is omitted in these patients.

SUMMARY:
Among ER+HER2- premenopausal patients with N1 who undergoes primary breast surgery, we will identify the patients with a genomic low risk using the multigene-assay (OncoFREE®).

In these, ovarian function suppression with endocrine therapies including either tamoxifen or aromatase-inhibitors will be administered for 5 years.

DETAILED DESCRIPTION:
* Among ER+HER2- premenopausal patients with N1 who undergoes primary breast surgery, we will identify the patients with a genomic low risk using the multigene-assay (OncoFREE®).
* In these, ovarian function suppression (OFS) with endocrine therapies including either tamoxifen or aromatase-inhibitors will be administered for 5 years.
* Either goserelin acetate or leuprorelin Acetate is allowed.
* These patients are able to choose bilateral salpingo-oophorectomy instead of OFS.
* Chemotherapy is omitted in these patients.

ELIGIBILITY:
Inclusion Criteria:

* ER+HER2- breast cancer
* Premenopausal and age <=50
* T1 or T2
* N1 including micrometastasis
* Genomic Low Risk by OncoFREE test® (1-20)

Exclusion Criteria:

* Postmenopausal women
* ER-negative breast cancer

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 418 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Distant recurrence-free survival | 5-years distant recurrence-free survival
  The interval between the date of primary surgery and the date of last censored, or distant recurrence or death of any cause

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | 5-years RFS
  The interval between the date of primary surgery and the date of last censored, or any type of recurrence or death of any cause
Invasive disease-free survival (iDFS) | 5-years iDFS
  The interval between the date of primary surgery and the date of last censored, or any type of invasive disease except thyroid cancer or death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Sung Gwe Ahn, M.D.,Ph.D., Principal Investigator — Gangnam Severance Hospital
Locations (2):
- South Korea (2):
  - Gangnam Severance Hospital, Seoul, Korea
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahn SG, Sim SH, Kang T, Kim EK, Lee JE, Moon HG, Ahn JH, Lim W, Youn HJ, Kim HA, Yoon CI, Kim J, Kang B, Park MH, Kang SH, Kim LS, Bae SJ, Kook Y, Lee KH, Lee HB, Han W, Park YH. Prospective Single-Arm Study of Endocrine Therapies With Ovarian Function Suppression in Premenopausal Node-Positive Early Breast Cancer Patients With Low Genomic Risk (INTERSTELLAR Trial, KBCSG-25). J Breast Cancer. 2026 Jan 30. doi: 10.4048/jbc.2025.0181. Online ahead of print. PMID 41612658